CLINICAL TRIAL: NCT03935009
Title: Learning Oral Hygiene Using Gamification: a Randomized Clinical Study
Brief Title: Learning Brushing Using Game Elements in Mobile Phones Apps
Acronym: GAMIFYBRUSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Maribor (Other)
Collaborators: Playbrush GmbH (Unknown); Flegis d.o.o. (Unknown); Middle-sized public primary school Videm pri Ptuju (Unknown)
Responsible Party: Principal Investigator, Nino Fijačko, Teaching assistant, University Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UM2019
Record Dates: First submitted 2019-04-16; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Oral Hygiene; Dental Plaque; Children, Only; Dental Devices, Home Care; Motivation; Learning
Keywords: Oral hygiene; Dental Plaque; Brushing; Flossing; Gamification; Game elements; Motivation; Education; Children; Parents
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual toothbrush with electric toothbrush N°1 (Active Comparator): Participants will receive manual toothbrush (Curaprox 5460 ultra soft, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Chomper Chums) and an electric toothbrush N°1 (Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Playbrush App) and will be instructed to use them for six weeks.
  Interventions: Behavioral: Manual toothbrush Curaprox 5460 ultra soft; Behavioral: Electric toothbrush Play Smart Brush N°1
- Manual toothbrush with electric toothbrush N°2 (Active Comparator): Participants will receive manual toothbrush (Curaprox 5460 ultra soft, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Chomper Chums) and an electric toothbrush N°2 (Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Utoothia) and will be instructed to use them for six weeks.
  Interventions: Behavioral: Manual toothbrush Curaprox 5460 ultra soft; Behavioral: Electric toothbrush Play Smart Brush N°2
- Electric toothbrush N°1 with electric toothbrush N°2 (Active Comparator): Participants will receive an electric toothbrush N°1 (Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Playbrush App) and an electric toothbrush N°2 (Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Utoothia) and will be instructed to use them for six weeks.
  Interventions: Behavioral: Electric toothbrush Play Smart Brush N°1; Behavioral: Electric toothbrush Play Smart Brush N°2

INTERVENTIONS:
Behavioral: Manual toothbrush Curaprox 5460 ultra soft — Soft manual toothbrush (Curaprox 5460 ultra soft) and Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Chomper Chumswill will be used to brush teeth.
  Arms: Manual toothbrush with electric toothbrush N°1; Manual toothbrush with electric toothbrush N°2
Behavioral: Electric toothbrush Play Smart Brush N°1 — Electric toothbrush (Play Smart Brush N°1) and Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Playbrush App will be used to brush teeth.
  Arms: Electric toothbrush N°1 with electric toothbrush N°2; Manual toothbrush with electric toothbrush N°1
Behavioral: Electric toothbrush Play Smart Brush N°2 — Electric toothbrush (Play Smart Brush N°2) and Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Utoothia will be used to brush teeth.
  Arms: Electric toothbrush N°1 with electric toothbrush N°2; Manual toothbrush with electric toothbrush N°2

SUMMARY:
The study aims to compare the efficacy of using gamification for oral hygiene in children at home environment.

DETAILED DESCRIPTION:
Subjects will be randomized into three groups:

1. The first group will receive a manual toothbrush Curaprox 5460 ultra soft, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Chomper Chums.
2. The second group will receive electric toothbrush Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Playbrush App.
3. The third group will receive electric toothbrush Playbrush Smart Sonic, Jordan Miracle Flossers floss, Curaprox toothpaste 1450 and mobile phone application Utoothia.

ELIGIBILITY:
Inclusion Criteria:

* Children with secondary dentition (not completed);
* Children age 10 years and above and don't have mental or physical disabilities;
* Children brushing teeth by themselves;
* Children using manual or electric toothbrush;
* Children using a mobile phone;

Exclusion Criteria:

* Children with the fixed orthodontic appliance;
* Children above 14 years;

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Control 1: Intrinsic motivation | Baseline
  The investigators will be using the Intrinsic Motivation Inventory (IMI) for measuring the participant intrinsic motivation (McAuley, Duncan, & Tammen, 1987). The IMI will have in total 37 items, measured on a 7-point scale.
Control 1: Oral hygiene index | Baseline
  The investigators will be using the Oral Hygiene Index (OHI) for measuring the participant debris Index (DI) and Calculus Index (CI) (Greene and Vermillion, 1960). Each index has a scale from 0 to 3. After the scores for DI and CI are recorded, the OHI (OHI range from 0 to 12) values are calculated. Higher the OHI, poorer is the oral hygiene of the participant.
Control 2: Intrinsic motivation | Two weeks after baseline
  The investigators will be using the Intrinsic Motivation Inventory (IMI) for measuring the participant intrinsic motivation (McAuley, Duncan, & Tammen, 1987). The IMI will have in total 37 items, measured on a 7-point scale.
Control 2: Oral hygiene index | Two weeks after baseline
  The investigators will be using the Oral Hygiene Index (OHI) for measuring the participant debris Index (DI) and Calculus Index (CI) (Greene and Vermillion, 1960). Each index has a scale from 0 to 3. After the scores for DI and CI are recorded, the OHI (OHI range from 0 to 12) values are calculated. Higher the OHI, poorer is the oral hygiene of the participant.
Control 3: Intrinsic motivation | Six weeks after baseline
  The investigators will be using the Intrinsic Motivation Inventory (IMI) for measuring the participant intrinsic motivation (McAuley, Duncan, & Tammen, 1987). The IMI will have in total 37 items, measured on a 7-point scale.
Control 3: Oral hygiene index | Six weeks after baseline
  The investigators will be using the Oral Hygiene Index (OHI) for measuring the participant debris Index (DI) and Calculus Index (CI) (Greene and Vermillion, 1960). Each index has a scale from 0 to 3. After the scores for DI and CI are recorded, the OHI (OHI range from 0 to 12) values are calculated. Higher the OHI, poorer is the oral hygiene of the participant.

SECONDARY OUTCOMES:
Oral hygiene knowledge of participants 1 | Baseline
  The investigators will use a questionnaire (Poutanen et al., 2007) about demographic factors and oral health-related knowledge attitudes, belief, and behavior to get information about the knowledge of participants oral health. Knowledge, attitudes, and beliefs are measured with 4-point Likert-scale questions; the alternatives were: strongly agree, partly agree, partly disagree, strongly disagree. Behaviors are measured with 7-point Likert-scale questions with alternatives that described the frequency of the behavior.
Oral hygiene knowledge of participants 2 | Six weeks after baseline
  The investigators will use a questionnaire (Poutanen et al., 2007) about oral health-related knowledge attitudes, belief, and behavior to get information about the knowledge of participants oral health. Knowledge, attitudes, and beliefs are measured with 4-point Likert-scale questions; the alternatives were: strongly agree, partly agree, partly disagree, strongly disagree. Behaviors are measured with 7-point Likert-scale questions with alternatives that described the frequency of the behavior.

OTHER OUTCOMES:
Indirect influence on oral hygiene of participants 1 | Baseline
  The investigators will use a combination of a different questionnaire from research (D'Cruz & Aradhya, 2012; de Silva-Sanigorski et al., 2013; Ramesh Kumar et al., 2013; Eden et al., 2018) about oral health to get information about the indirect influence on the oral hygiene of participants.
Indirect influence on oral hygiene of participants 2 | Six weeks after baseline
  The investigators will use a combination of a different questionnaire from research (D'Cruz & Aradhya, 2012; de Silva-Sanigorski et al., 2013; Ramesh Kumar et al., 2013; Eden et al., 2018) about oral health to get information about the indirect influence on the oral hygiene of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Nino Fijacko, Study Chair — University Maribor
Locations (2):
- Slovenia (2):
  - University Maribor, Maribor
  - University of Maribor Faculty of health sciences, Maribor

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and all data will be part of the published article in the journal.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publishing an article in the journal.
Access Criteria: No special criteria.
URL: https://sites.google.com/view/zobek

REFERENCES:
- [Background] Acharya S, Goyal A, Utreja AK, Mohanty U. Effect of three different motivational techniques on oral hygiene and gingival health of patients undergoing multibracketed orthodontics. Angle Orthod. 2011 Sep;81(5):884-8. doi: 10.2319/112210-680.1. Epub 2011 May 25. PMID 21612316
- [Background] Kotha SB, Alabdulaali RA, Dahy WT, Alkhaibari YR, Albaraki ASM, Alghanim AF. The Influence of Oral Health Knowledge on Parental Practices among the Saudi Parents of Children Aged 2-6 Years in Riyadh City, Saudi Arabia. J Int Soc Prev Community Dent. 2018 Nov-Dec;8(6):565-571. doi: 10.4103/jispcd.JISPCD_341_18. Epub 2018 Nov 29. PMID 30596050
- [Background] Marshman Z, Ahern SM, McEachan RRC, Rogers HJ, Gray-Burrows KA, Day PF. Parents' Experiences of Toothbrushing with Children: A Qualitative Study. JDR Clin Trans Res. 2016 Jul;1(2):122-130. doi: 10.1177/2380084416647727. Epub 2016 Apr 26. PMID 28879241
- [Background] Harnacke D, Mitter S, Lehner M, Munzert J, Deinzer R. Improving oral hygiene skills by computer-based training: a randomized controlled comparison of the modified Bass and the Fones techniques. PLoS One. 2012;7(5):e37072. doi: 10.1371/journal.pone.0037072. Epub 2012 May 21. PMID 22629353
- [Background] Credé M, Phillips LA. A meta-analytic review of the Motivated Strategies for Learning Questionnaire. Learning and individual differences 21(4): 337-46, 2011.
- [Background] Pan N, Cai L, Xu C, Guan H, Jin Y. Oral health knowledge, behaviors and parental practices among rural-urban migrant children in Guangzhou: a follow-up study. BMC Oral Health. 2017 Jun 7;17(1):97. doi: 10.1186/s12903-017-0385-2. PMID 28592239
- [Background] Soltani R, Ali Eslami A, Mahaki B, Alipoor M, Sharifirad G. Do maternal oral health-related self-efficacy and knowledge influence oral hygiene behavior of their children?. International Journal of Pediatrics 4(7): 2035-42, 2016.
- [Background] Wilson A, Brega AG, Batliner TS, Henderson W, Campagna EJ, Fehringer K, Gallegos J, Daniels D, Albino J. Assessment of parental oral health knowledge and behaviors among American Indians of a Northern Plains tribe. J Public Health Dent. 2014 Spring;74(2):159-67. doi: 10.1111/jphd.12040. Epub 2013 Oct 9. PMID 24117628
- [Background] Wilson M, Morgan M. A survey of children's toothbrushing habits in Wales: Are parents following the guidelines?. Journal of Health Visiting 4(2):95-9, 2016.
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Poutanen R, Lahti S, Seppa L, Tolvanen M, Hausen H. Oral health-related knowledge, attitudes, behavior, and family characteristics among Finnish schoolchildren with and without active initial caries lesions. Acta Odontol Scand. 2007 Apr;65(2):87-96. doi: 10.1080/00016350601058077. PMID 17453426
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Background] D'Cruz AM, Aradhya S. Impact of oral health education on oral hygiene knowledge, practices, plaque control and gingival health of 13- to 15-year-old school children in Bangalore city. Int J Dent Hyg. 2013 May;11(2):126-33. doi: 10.1111/j.1601-5037.2012.00563.x. Epub 2012 Jun 30. PMID 22747831
- [Background] de Silva-Sanigorski A, Ashbolt R, Green J, Calache H, Keith B, Riggs E, Waters E. Parental self-efficacy and oral health-related knowledge are associated with parent and child oral health behaviors and self-reported oral health status. Community Dent Oral Epidemiol. 2013 Aug;41(4):345-52. doi: 10.1111/cdoe.12019. Epub 2012 Nov 17. PMID 23157162
- [Background] Eden E, Akyildiz M, Sonmez I. Comparison of Two School-Based Oral Health Education Programs in 9-Year-Old Children. Int Q Community Health Educ. 2019 Apr;39(3):189-196. doi: 10.1177/0272684X18819980. Epub 2018 Dec 21. PMID 30577724
- [Background] Kumar SR, Narayanan MA, Jayanthi D. Comparison of oral hygiene status before and after health education among 12-18-year-old patients. Journal of Indian Association of Public Health Dentistry 14(2):121, 2016.
- See also: Official questionnaire about intrinsic motivation which will be used for measure motivation for learning oral hygiene. — https://gih.instructure.com/files/2040/download?download_frd=1